CLINICAL TRIAL: NCT07120217
Title: Breast Cancer Risk Investigation in Grown-up Hodgkin Lymphoma Patients Treated With MBVD.
Brief Title: Breast Cancer Risk Investigation in Grown-up Hodgkin Lymphoma Patients Treated With MBVD. Multicenter Retrospective Study on ≥200 Adult Female HL Patients Treated With ≥1 MBVD Cycle (NPLD, Bleomycin, Vinblastine, Dacarbazine). It Investigates Breast Cancer Incidence Post-treatment.
Acronym: BRIGHT-MBVD
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Marco Picardi, Full Professor, Federico II University
Other Study IDs: BRIGHT-MBVD
Record Dates: First submitted 2025-08-01; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Hodgkin Disease; Breast Cancer; Liposomal Doxorubicin
Keywords: non pegilated liposomal doxorubicin
MeSH Terms: conditions — Hodgkin Disease; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This is a multicenter retrospective cohort study conducted at the Hematology Unit of the University of Naples Federico II and the Hematology Department of AORN Cardarelli, Naples, Italy. The study investigates the incidence of breast cancer in adult female patients (aged ≥18 years) diagnosed with classical Hodgkin lymphoma (HL) and treated with at least one cycle of MBVD chemotherapy (liposomal doxorubicin [NPLD], bleomycin, vinblastine, dacarbazine). All diagnoses are made according to the WHO Classification of Lymphoid Neoplasms.

Ethics and Consent:

The study will be conducted in accordance with the principles of the Declaration of Helsinki. All participants will provide written informed consent for data collection and analysis. Approval by the local Institutional Ethics Committee will be obtained prior to data collection.

Study Objectives:

The primary aim is to evaluate the incidence of secondary breast cancer in female HL survivors treated with NPLD-based chemotherapy (MBVD). The potential association between NPLD and breast cancer risk has not been comprehensively studied in adult HL survivors. This study seeks to address this gap by analyzing long-term outcomes in a well-defined patient population. The target sample size is a minimum of 200 patients.

Data Collection and Study Timeline:

Eligible patients undergoing hematological follow-up at the two participating institutions will be invited to participate. Upon consent, data will be extracted from patient records and entered into standardized case report forms (CRFs). The expected duration of data collection is approximately 2 months. The observational window spans from January 2000 to July 2025.

Therapeutic Regimen:

All patients received at least one cycle of the MBVD regimen, which includes:

NPLD (Myocet™) 25 mg/m² IV on days 1 and 15, every 28 days

Bleomycin 10 mg/m² IV on days 1 and 15, every 28 days

Vinblastine 6 mg/m² IV on days 1 and 15, every 28 days

Dacarbazine 375 mg/m² IV on days 1 and 15, every 28 days

The cumulative NPLD dose remained well below the cardiotoxicity threshold of 785 mg/m². End-of-treatment evaluation included a total-body FDG-PET scan.

Radiotherapy and Supportive Therapy:

Consolidative radiotherapy (30 Gy) was administered to patients with bulky disease at diagnosis (defined as nodal mass >5 cm). All patients received standard antimicrobial prophylaxis:

Oral trimethoprim-sulfamethoxazole 960 mg (160+800 mg) twice weekly

Oral acyclovir 800 mg daily from the first day of chemotherapy until one month after the last cycle Additional supportive treatments were administered at the discretion of the treating physician.

Follow-Up and Imaging:

FDG-PET/CT was performed for staging, at the end of therapy, and subsequently every 3-6 months. PET results were interpreted using the Deauville Score (DS) and Lugano criteria:

Negative PET: DS ≤3

Positive PET: DS 4 or 5

Cardiac Monitoring:

All patients underwent comprehensive cardiac assessment, including baseline, interim, and end-of-treatment (EoT) 2D echocardiography and speckle-tracking echocardiography (STE). Additional cardiac evaluations were performed within six months of completing antineoplastic therapy.

Expected Outcomes:

The study aims to assess the long-term breast cancer risk associated with NPLD-containing regimens in HL patients, a population in which long-term toxicities remain under-investigated. The results may inform future recommendations on post-treatment surveillance and guide oncologic decision-making in young adult HL patients.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed diagnosis of classical Hodgkin lymphoma (HL)

Female sex

Age ≥18 years at the time of diagnosis

Treatment with ≥1 cycle of MBVD chemotherapy regimen

ECOG Performance Status (PS) 0-3

HIV negative status

Signed informed consent to participate in the study and for data analysis

Exclusion Criteria:

Incomplete or inadequate breast cancer surveillance work-up (i.e., lacking appropriate breast imaging such as ultrasound, mammography, MRI, or cytologic/histologic assessment if clinically indicated)

Last HL-related therapy (of any line) received within 5 years from the last hematological follow-up visit

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Female patients will be identified from the hematology outpatient databases of two tertiary referral centers in Naples, Italy: the Hematology Unit at the University Hospital Federico II and the Hematology Department at AORN Cardarelli. Participants are long-term Hodgkin lymphoma survivors who received follow-up care at these institutions between January 2000 and July 2025.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-01-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Breast Cancer Following MBVD Therapy | from 1 January 2000 to 1 July 2025
  The primary endpoint is the cumulative incidence of breast cancer among adult female Hodgkin lymphoma survivors treated with MBVD (liposomal doxorubicin, bleomycin, vinblastine, dacarbazine). Breast cancer cases will be confirmed by histologic or cytologic examination and classified according to international oncologic standards.